CLINICAL TRIAL: NCT01780961
Title: Prospective Collection of Health Information and Biospecimens in Esophageal Cancer
Brief Title: Esophageal Cancer Tissue Banking
Acronym: ESBX
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201101765
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Cancer; ESBX
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — peripheral blood and Esophageal Tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
To create an esophageal cancer biospecimen repository that will collect, annotate, store and distribute human esophageal cancer biospecimens in a manner that embraces the highest ethical standards of human subject's research, that conforms to the best practices of biorepository science and that furthers basic, translational and clinical research in the understanding diagnosis and treatment of this disease.

DETAILED DESCRIPTION:
Prospective databases have contributed substantially to the advancement of clinical medicine and surgery. Examples of contributions from databases include an improved understanding of the treatment and outcome for rare pathologies, the long term outcomes, and incidence of uncommon complications from more common disease, and the repercussions of infrequently performed complex procedures. (1-3) Problems identified by database review have led to improvements in patient care and have guided the planning of numerous prospective studies. The value of these databases incrementally increases with the number of patients enrolled and with the length of time the databases have been maintained. Recently databases have been used to create and test nomograms, which are increasingly being implemented to further refine patient prognosis and to stratify patients for clinical trials. (4) We anticipate that a prospective database will become more valuable as we look to the future. Increasingly, molecular markers are identified which are thought to be important to patient outcome or treatment response. When linked to pathologic tissues, clinical databases can be used as the initial test of these newly identified markers and to determine which warrant an independent prospective review. An independent prospective analysis performed for each marker is costly and time consuming. A prospective database is more comprehensive, accurate, and ultimately less time consuming than retrospective review for testing each set of markers as novel questions arise.

This study will augment a prospective database of patients with esophageal cancer who undergo investigation and /or surgery at Washington University School of Medicine. This database will be periodically updated from the patient records and the computerized medical record as patients continue routine follow-up care. These data will be used to address questions regarding treatment and/or disease-specific outcomes.

In addition, we seek to acquire, store and analyze tissue and blood samples on these patients. Samples will be processed and stored at the Tissue Procurement Facility of Washington University School of Medicine. We will be using this material to support ongoing efforts to identify serum markers with applications for early diagnosis, prognosis or treatment efficacy. Markers identified will be linked to the clinical outcomes data as captured in the database. Using the database, we will be able to link patient and treatment outcomes to analyses performed on previously collected pathologic specimens or research specimens and correlate these results with the patients' treatment response and outcome in a time efficient and cost effective way.

The incidence of esophageal adenocarcinoma is on the rise. This has been a trend that has been noted over the last decade and has gone hand in hand with a decrease in the incidence of esophageal squamous cell carcinoma. Overall the number of patients with esophageal cancer being diagnosed annually in the United States is steadily increasing. Esophageal cancer afflicts approximately 19,000 patients annually in the United States. Broadly speaking, esophageal cancer can be diagnosed at an early stage where there is no metastatic disease in distant organs or at a relatively advanced stage when there is evidence of metastatic disease in distant organs. Unfortunately patients with metastatic disease can receive only palliative therapy and survival is quite limited. Stage I - III esophageal cancer is often treated either by primary surgery or by a combination of preoperative or postoperative chemoradiation therapy along with surgical resection. For stage I esophageal cancer, surgical resection usually suffices and patients have upwards of 70-80% five year survival. For patients with stage III esophageal cancer, the patients usually undergo induction chemoradiation therapy followed by surgical resection. Induction chemoradiation usually involves two cycles of % Fluorouracil and cisplatin with 5040 Gy of external beam radiation therapy. This aspect of treatment has been well standardized (5). For stage II esophageal cancer, surgery forms the backbone of therapy, however, there is no clear consensus among treating physicians about the efficacy and role of chemoradiation therapy in these patients.

In patients who undergo chemoradiation therapy prior to surgery for esophageal cancer, it is noted that 15-30% of patients have had a complete pathologic response to therapy. Thus no tumor is detected in the resected specimen in these patients. Therefore, theoretically, these patients have undergone an unnecessary resection. There is currently no way to predict which patients would have had a pathologic response short of resecting the esophagus and thus exposing the patients to the significant morbidity and mortality associated with this major operation.

The most significant impact of next-generation sequencing on cancer genomics has been the ability to re-sequence, analyze and compare the matched tumor and normal genomes of a single patient. With the significantly reduced cost of sequencing and tremendously enhanced throughput, it is now within the realm of possibility to sequence multiple patient samples of a given cancer type. Genomic analyses over the last few years, with significant contributions from our own Genome Center at the Washington University in St. Louis, (6-7) have led to significant advances in understanding the behavior of certain tumors including leukemias and glioblastoma. Specifically, in acute leukemias, our center has shown that certain genotypes of the tumor predict favorable or unfavorable outcomes in the patients analyzed. These findings now have been replicated in at least 3 independent studies of separate AML cohorts. Our goal with this project would be to develop an understanding of the genomic profile of esophageal carcinomas and changes with treatment. Furthermore with availability of tissue both before and after chemoradiation therapy, we would be able to identify changes in the genome of the malignancy with induction therapy. Also with resection specimens we will be able to identify which patients have had a significant response to therapy (including complete pathologic response) and others who have not had a significant response to therapy or have had progressive disease despite therapy. This may help us in identifying genomic features of the spectrum of esophageal carcinomas that predict response to therapy after having had the chance to longitudinally study the disease or the clinical course of the patients. Specifically this would be achieved by obtaining tissue specimens from the malignancy prior to any therapy at the time of the initial diagnosis or initial endoscopy for these patients. Subsequently the patients would undergo routine therapy which would be based upon their clinical stage of disease. Eventually when patients come back for their definitive resection, we would be able to access the pathologic profile to assess response to induction therapy and also to study the genomic profile of the tumor tissue after induction therapy.

A prospective database which would be maintained in the Division of Cardiothoracic Surgery would be able to link clinical outcomes to processed tissues (pathologic specimens, research specimens and plasma) enabling higher level correlation studies to be performed. Proper use of such a resource will aid considerably in our ability to advance our field and care for our future patients with esophageal cancer.

Our eventual aim with the analyses of the genome of esophageal cancer would be to identify a patient population that has a complete pathologic response to chemoradiation therapy for carcinomas of the esophagus. We will be able to identify genomic differences, if any, between such tumors and other tumors where there is only a partial response/no response/progressive disease with induction chemoradiation therapy. If analyses are sufficiently predictive and efficiently dichotomize patients into these categories based upon genomic profiles, this can be the lead groundwork for a clinical trial where patients with certain specific genomic profiles would be treated only with chemoradiation therapy for carcinomas of the esophagus, thus precluding unnecessary surgery with its significant attendant morbidity and mortality. As we already know, about 15-30% of patients undergoing induction chemoradiation therapy clinically fall into such a category. The well known morbidity of an esophagectomy includes significant pulmonary problems, anastomotic leaks, cardiovascular problems, chyle leak, venous thromboses, amongst other major problems. The rate of morbidity after an esophagectomy varies from 20-40%. Also there is 3-14 % risk of mortality from esophagectomy. (8-9) Therefore, a tool that can effectively predict which patients do not require an esophagectomy for treatment of carcinomas of the esophagus would be extremely useful clinically.

ELIGIBILITY:
Inclusion Criteria:

* Adults with known or suspected esophageal cancer who are willing and able to give written informed consent for biospecimen collections.
* Age ≥ 18 years
* Must be willing and able to sign an informed consent document

Exclusion Criteria:

* Pediatric patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be identified by participating staff in the clinics of the surgical oncology or medical oncology clinics, and patients referred to the endoscopy center, and provided information about the biorepository.
Sampling Method: Probability Sample
Enrollment: 311 (Actual)
Dates: Start 2011-01-25 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Prospective Database | five years
  A prospective database which would be maintained in the Division of Cardiothoracic Surgery would be able to link clinical outcomes to processed tissues (pathologic specimens, research specimens and plasma) enabling higher level correlation studies to be performed. Proper use of such a resource will aid considerably in our ability to advance our field and care for our future patients with esophageal cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Edwards FH. The STS database at 20 years: a tribute to Dr Richard E. Clark. Ann Thorac Surg. 2010 Jan;89(1):9-10. doi: 10.1016/j.athoracsur.2009.11.028. No abstract available. PMID 20103196
- [Background] Ferguson TB Jr, Dziuban SW Jr, Edwards FH, Eiken MC, Shroyer AL, Pairolero PC, Anderson RP, Grover FL. The STS National Database: current changes and challenges for the new millennium. Committee to Establish a National Database in Cardiothoracic Surgery, The Society of Thoracic Surgeons. Ann Thorac Surg. 2000 Mar;69(3):680-91. doi: 10.1016/s0003-4975(99)01538-6. PMID 10750744